CLINICAL TRIAL: NCT01184417
Title: Phenobarbital Versus Placebo for Acute Alcohol Withdrawal
Brief Title: Phenobarbital for Acute Alcohol Withdrawal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonathan Rosenson (Other)
Collaborators: Alameda County Medical Center (Other)
Responsible Party: Sponsor-Investigator, Jonathan Rosenson, Jonathan Rosenson MD, Alameda County Medical Center
Organization: Alameda County Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AlamedaCountyMC
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Results first posted 2012-03-09 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Alcohol Withdrawal
MeSH Terms: interventions — Phenobarbital; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phenobarbital group (Active Comparator): 10 mg/kg IV phenobarbital in 100 ml saline
  Interventions: Drug: 10 mg/kg IV phenobarbital in 100 ml saline
- Placebo group (Placebo Comparator): 100 ml saline
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 10 mg/kg IV phenobarbital in 100 ml saline — 10 mg/kg IV phenobarbital in 100 ml saline
  Arms: Phenobarbital group
Drug: placebo — 100 m l saline
  Arms: Placebo group

SUMMARY:
Intravenous phenobarbital in combination with a symptom-guided standardized lorazepam-based alcohol withdrawal protocol will be associated with decreased need for ICU admission, continuous lorazepam infusion and will not be associated with increased adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Need for admission to hospital for acute alcohol withdrawal

Exclusion Criteria:

* allergy to phenobarbital, lorazepam, age<18 or >65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alameda County Medical Center, Oakland, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phenobarbital Group | Placebo Group
Started | 51 | 51
Completed | 51 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenobarbital Group | Placebo Group | Total
Number analyzed (Participants) | 51 | 51 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 51 | 102
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46 (12) | 48 (17) | 47 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 45 | 91
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 51 | 51 | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Requiring Continuous Lorazepam Infusion
Description: All study patients are placed on the standardized institutional alcohol withdrawal protocol and receive boluses of lorazepam (1, 2 or 4 mg IV) based on their acute alcohol withdrawal score (AAWS), adminstered serially up to every 15 minutes. Patients who are refractory to the maximum dose of lorazepam allowed by the protocol (up to 4mg lorazepam IV q 15 mins)are placed on a continuous IV lorazepam infusion (or "lorazepam drip"). Thus, continuous lorazepam infusion is a "yes or no" variable (i.e. continuous infusion, or not).
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Phenobarbital Group | Placebo Group
Number analyzed (Participants) | 51 | 51
participants | 2 | 16

2. Primary Outcome: Percentage of Patients Requiring ICU Admission
Description: admission to intensive care unit
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Phenobarbital Group | Placebo Group
Number analyzed (Participants) | 51 | 51
percentage of participants | 8 [4 to 32] | 25 [4 to 32]
Statistical Analysis 1: Comparison: Phenobarbital Group vs Placebo Group; Test type: Superiority or Other; Mean Difference (Final Values) = 17, 95% CI 2-sided [4 to 32]

3. Primary Outcome: Total Lorazepam Required Per Patient Per Admission
Description: How much total lorazepam did each study patient receive from inital presentation in the Emergency Department through their discharge from the hospital, in milligrams.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Phenobarbital Group | Placebo Group
Number analyzed (Participants) | 51 | 51
milligrams | 26 (45) [7 to 49] | 49 (37) [7 to 49]
Statistical Analysis 1: Comparison: Phenobarbital Group vs Placebo Group; Test type: Superiority or Other; Mean Difference (Final Values) = 23, 95% CI 2-sided [4 to 49]

4. Secondary Outcome: Length of Stay
Description: hospital LOS, per patient, in hours from admission to discharge
Time Frame: 1 year
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Phenobarbital Group | Placebo Group
Number analyzed (Participants) | 51 | 51
hours | 76 [54 to 114] | 118 [47 to 190]
Statistical Analysis 1: Comparison: Phenobarbital Group vs Placebo Group; Test type: Superiority or Other; Mean Difference (Final Values) = 42, 95% CI 2-sided [-4 to 82]

5. Secondary Outcome: Number of Patients Requiring Endotracheal Intubation as a Measure of Safety and Tolerability
Description: The outome answeres the question "Did the study patient require endotracheal intubation, or not". This outcome investigates if the phenobarbital intervention is associted with increased incidence of respiratory depression and subsequent increased need for intubation.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Phenobarbital Group | Placebo Group
Number analyzed (Participants) | 51 | 51
participants | 0 | 0

6. Secondary Outcome: Percentage of Patients Requiring a Bedside Sitter as a Measure of Safety and Tolerability
Description: Did the study patient require a Licensed Vocational Nurse (LVN) or other hospital staff to serve as a "bedside sitter" to observe the patient and provide additional safety supervision during any portion of their hospitalization.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Phenobarbital Group | Placebo Group
Number analyzed (Participants) | 51 | 51
percentage of participants | 28 [-11 to 23] | 22 [-11 to 23]
Statistical Analysis 1: Comparison: Phenobarbital Group vs Placebo Group; Test type: Superiority or Other; Mean Difference (Final Values) = 6, 95% CI 2-sided [-11 to 23]

7. Secondary Outcome: Number of Study Patients With Seizure as a Measure of Safety and Tolerability
Description: Did the study patient have a witnessed seizure during their hospitaliztion (yes/no).
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Phenobarbital Group | Placebo Group
Number analyzed (Participants) | 51 | 51
participants | 1 | 2

8. Secondary Outcome: Number of Study Patients With Mortality as a Measure of Safety and Tolerability
Description: mortality in study patients
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Phenobarbital Group | Placebo Group
Number analyzed (Participants) | 51 | 51
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Phenobarbital Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/51
Other Adverse Events (participants affected / at risk) | 0/51 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes